CLINICAL TRIAL: NCT07188259
Title: Prevalence and Impact of Heavy Menstrual Bleeding Among Female Students in Assiut University, Egypt
Brief Title: Prevalence and Impact on Quality of Life, Academic Performance, and Blood Indices of Heavy Menstrual Bleeding Among Female Students in Assiut University, Egypt
Acronym: menorrhagia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Ismail Mohamed, Principal Investigator, Assiut University
Other Study IDs: PIHMBFSAUE
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Heavy menstrual bleeding positive group: After using the SAMANTA scale, if we find a score of 3 or more, this will be:
  Heavy menstrual bleeding positive group
- Heavy menstrual bleeding negative group: After using the SAMANTA scale, if we find a score less than 3, this will be:
  Heavy menstrual bleeding negative group

SUMMARY:
The cause of menstrual disorders is unknown because many female students, embarrassed or unsure of what is "normal," never seek care. In young females, abnormal uterine bleeding is usually functional-reflecting immaturity or dysregulation of the hypothalamic-pituitary-ovarian axis, anovulatory cycles, or inherited bleeding disorders-while serious structural pathology is rare. Nevertheless, early bleeding can be the first sign of conditions such as polycystic-ovary syndrome, endometriosis, or von Willebrand disease. It is the primary source of iron-deficiency anemia in females before marriage, leading to chronic fatigue, diminished academic performance, and lower exam results.

A sectional study will be performed using a semi-structured questionnaire to assess the presence of HMB using the SAMANTA scale after its Arabic validation, and also evaluate the effect of HMB on quality of life using the validated heavy menstrual bleeding scale and assess impact on academic performance finally both females with positive HMB or not will asked to do Complete blood count (CBC), serum ferritin and coagulation profile.

ELIGIBILITY:
Inclusion Criteria:

1- Female students of Assiut University.

Exclusion Criteria:

1. Females known to have chronic anemia or hemolytic anemia by history
2. Females on anticoagulation treatment.
3. Females known to have coagulopathy.
4. Females with any chronic condition (diabetes mellitus, liver diseases, etc.) in the previous 12 months were excluded from participation in this study.
5. Females with a history of prior pregnancy (gravidity ≥1), regardless of outcome (live birth, miscarriage, abortion, or ectopic).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Female Students in Assiut University, Egypt who accepted to share in the study
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
the prevalence of heavy menstrual bleeding (HMB) | through study completion, an average of 6 months to 1 year.
  to estimate the prevalence of heavy menstrual bleeding (HMB) among Assiut university female students.

SECONDARY OUTCOMES:
impact of heavy menstrual bleeding (HMB) on participants' quality of life and academic performance. | through study completion, an average of 6 months to 1 year
  To evaluate the impact of heavy menstrual bleeding (HMB) on participants' quality of life and academic performance.
Hematologic (CBC indices, serum ferritin and coagulation profile) between participants | within 2 months after questionnaire
  Compare hematologic (CBC indices, serum ferritin and coagulation profile) between participants with HMB and partcipants without HMB.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University,, Asyut, Egypt

REFERENCES:
- [Background] Nwagha TU, Okoye HC, Ugwu AO, Ugwu EO. Clinical screening for menorrhagia and other bleeding symptoms in Nigerian women. Ann Afr Med. 2021 Apr-Jun;20(2):111-115. doi: 10.4103/aam.aam_26_20. PMID 34213477
- [Background] Sinharoy SS, Chery L, Patrick M, Conrad A, Ramaswamy A, Stephen A, Chipungu J, Reddy YM, Doma R, Pasricha SR, Ahmed T, Chiwala CB, Chakraborti N, Caruso BA. Prevalence of heavy menstrual bleeding and associations with physical health and wellbeing in low-income and middle-income countries: a multinational cross-sectional study. Lancet Glob Health. 2023 Nov;11(11):e1775-e1784. doi: 10.1016/S2214-109X(23)00416-3. Epub 2023 Oct 3. PMID 37802092